CLINICAL TRIAL: NCT03799991
Title: Vestibular Therapy in Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00273752; R01AG065259 (NIH)
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Vestibular Diseases; Vestibular Disorder; Alzheimer Disease
MeSH Terms: conditions — Vestibular Diseases; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular therapy (Experimental): Vestibular therapy (Vestibular physical therapy) entails an 8-week course of exercises delivered by a physical therapist designed to improve vestibular function.
  Interventions: Behavioral: Vestibular physical therapy
- Active control (Active Comparator): The active control regimen consists of eye movement exercises (e.g. smooth pursuit eye movements) and also general conditioning exercises (e.g. range of motion exercises, lifting light weights with the arms and legs). This regimen is "vestibular neutral" in that head movements which specifically challenge the vestibular system are avoided.
  Interventions: Behavioral: Active control

INTERVENTIONS:
Behavioral: Vestibular physical therapy — Vestibular therapy is a set of exercises delivered by a physical therapist involving head movements. The therapy is delivered over a course of 8 weeks.
  Arms: Vestibular therapy
Behavioral: Active control — Strength and flexibility exercises that do not involve head movements.
  Arms: Active control

SUMMARY:
Nearly 2 out of 3 patients with Alzheimer's disease (AD) experience problems with balance and mobility, which places such patients at increased risk of falling. The vestibular (inner ear balance) system plays an important role in balance stability, and vestibular therapy (VT) is well-known to improve balance function in healthy older adults. In this study, the investigators will conduct a first-in-kind randomized clinical trial to evaluate whether vestibular therapy improves reduces falls in patients with AD, in whom this treatment has never been studied.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD based on the National Institute on Aging-Alzheimer Association 2011 criteria that is mild-moderate (CDR=0.5-2).
* Age ≥ 60 years.
* Vestibular loss defined as bilaterally impaired vestibular responses (semicircular canal or otolith responses).
* Able to participate in study procedures including vestibular physiologic testing, balance and gait assessment, neurocognitive testing, and VT or active control.
* Able to give informed consent, as further detailed in the Human Subjects section. The investigators anticipate that individuals who are too impaired to provide informed consent would also not be able to effectively participate in VT or active control.
* Presence of a caregiver, defined as an individual who spends at least 10 hours per week with the patient. The caregiver must be able to participate in study procedures, specifically the text-messaging system. Both the VT and active control involve 8 weeks of once weekly visits and daily home exercises, and the investigators believe a caregiver would increase the likelihood of successful completion of either therapy.

Exclusion Criteria:

* Diagnosis of severe AD (CDR≥3).
* Diagnosis of mild cognitive impairment or diagnosis of non-AD dementia, for example Parkinson's disease dementia, Dementia with Lewy Bodies, vascular dementia, fronto-temporal dementia, and primary progressive aphasia.
* Deemed unable to participate in study procedures and VT or active control, (e.g. patients with significant medical comorbidities, excessive agitation, or use of mobility aids such as a cane or walker.)
* Use of daily vestibular suppressant medications, specifically anti-histamines and benzodiazepines, as this can alter the response to VT.
* Lack of availability to participate in 8 weeks of VT or active control.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2027-08-26 (Estimated); Study Completion 2027-08-26 (Estimated)

PRIMARY OUTCOMES:
Number of participant falls | 1 year
  Incidence of falls over a 1-year follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Agrawal, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yesantharao LV, Rosenberg P, Oh E, Leoutsakos J, Munro CA, Agrawal Y. Vestibular therapy to reduce falls in people with Alzheimer's disease: study protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2022 Aug 2;8(1):167. doi: 10.1186/s40814-022-01133-w. PMID 35918757